CLINICAL TRIAL: NCT05261516
Title: Interaction Between Intravenous Magnesium Sulfate and Volatile Anesthetics Compared to Propofol. A Three-center Prospective Randomized Single-blinded Electrophysiological Study
Brief Title: Interaction of Volatile Anesthetics With Magnesium
Acronym: Volmag
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Christoph Czarnetzki (Other)
Collaborators: Centre Hospitalier du Centre du Valais (Other); Ospedale Regionale di Lugano (Other)
Responsible Party: Sponsor-Investigator, Christoph Czarnetzki, Consultant, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2019-02104/CE3541
Record Dates: First submitted 2020-04-09; First posted 2022-03-02 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Neuromuscular Blockade
Keywords: Magnesium; Volatiles anesthetics; Neuromuscular transmission
MeSH Terms: interventions — Magnesium Sulfate

STUDY DESIGN:
Intervention Model Description: This study is a three centers prospective randomized, electrophysiological, single blinded study that will include 96 patients allocated to one of four arms: one arm with propofol anesthesia and three arms with volatile anesthetics (one arm with isoflurane, one with sevoflurane and one with desflurane). Each arm will have 24 patients.
Who Masked: Participant
Masking Description: For practical reasons it is impossible to blind the investigator who conducts the anesthesia. However, the parameters of neuromuscular block are standardized, and study outcomes will be evaluated using the data stored and displayed in theTetraGraph Viewer software. All neuromuscular measurements of the study outcomes are reproducible and objective.
  In contrast, the investigator evaluating the patient in the postanesthetic care unit and for the 24 h postoperative visit will be blinded to the study group allocation.
  The patient will also be blinded to the study group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Propofol (Active Comparator): In all patients 3 minutes before induction sufentanil 0.2 mcg/kg or fentanyl 2 mcg/kg will be given.
  In patients in the propofol group, anesthesia will be induced and maintained with a total intravenous anesthesia pump following the model of Schnider et al, at a targeted effect-site concentration of 4 +/- 1 mcg/ml.
  In patients in all groups, after induction of anesthesia and loss of consciousness, a laryngeal mask airway will be inserted. The TetraGraph device will be calibrated. Once general anesthesia is established, a blood sample will be taken to measure serum magnesium and calcium levels. This blood sample will be analysed in the certified laboratory of each participating hospital.
  Interventions: Drug: Magnesium Sulfate
- Isoflurane (Experimental): In all patients 3 minutes before induction sufentanil 0.2 mcg/kg or fentanyl 2 mcg/kg will be given. After induction of anesthesia and loss of consciousness, a laryngeal mask airway will be inserted. The TetraGraph device will be calibrated. Once general anesthesia is established, a blood sample will be taken to measure serum magnesium and calcium levels. This blood sample will be analysed in the certified laboratory of each participating hospital.
  The anesthesia will be maintained with the agent specified by randomization: isoflurane in this group.
  Interventions: Drug: Magnesium Sulfate
- Desflurane (Experimental): In all patients 3 minutes before induction sufentanil 0.2 mcg/kg or fentanyl 2 mcg/kg will be given. After induction of anesthesia and loss of consciousness, a laryngeal mask airway will be inserted. The TetraGraph device will be calibrated. Once general anesthesia is established, a blood sample will be taken to measure serum magnesium and calcium levels. This blood sample will be analysed in the certified laboratory of each participating hospital.
  The anesthesia will be maintained with the agent specified by randomization: desflurane in this group.
  Interventions: Drug: Magnesium Sulfate
- Sevoflurane (Experimental): In all patients 3 minutes before induction sufentanil 0.2 mcg/kg or fentanyl 2 mcg/kg will be given. After induction of anesthesia and loss of consciousness, a laryngeal mask airway will be inserted. The TetraGraph device will be calibrated. Once general anesthesia is established, a blood sample will be taken to measure serum magnesium and calcium levels. This blood sample will be analysed in the certified laboratory of each participating hospital.
  The anesthesia will be maintained with the agent specified by randomization: sevoflurane in this group.
  Interventions: Drug: Magnesium Sulfate

INTERVENTIONS:
Drug: Magnesium Sulfate — The experimental intervention is the injection of magnesium sulfate. This will be done as soon as TetraGraph calibration is done and neuromuscular measurements are stable. Each patient will receive 60 mg/kg of magnesium sulfate as an intravenous perfusion over 5 minutes. Vital signs before, during and after the perfusion will be taken and documented.

SUMMARY:
Magnesium and volatiles anesthetics both have an effect on the neuromuscular transmission. The primary objective of the study is to quantify the effect of a perfusion of intravenous magnesium on neuromuscular transmission measured by electromyography device TetraGraph device in patients undergoing general anesthesia with volatile anesthetics (desflurane, sevoflurane and isoflurane) as compared to intravenous anesthesia with propofol.

DETAILED DESCRIPTION:
Magnesium sulfate is regularly used during anesthesia, for instance for the reduction of postoperative pain. It reduces the liberation of acetylcholine at the neuromuscular junction. At high plasma concentrations it can induce muscle weakness, flaccid paralysis and in cases of intoxication lead to respiratory arrest. It enhances the effect of muscle relaxants.

Volatiles anesthetics influence neuromuscular transmission. They inhibit postsynaptic nicotinic acetylcholine receptors by causing open channel block, receptor desensitization and reducing exocytosis from pre-synaptic vesicles at the neuromuscular junction. The ranking order of these effects of volatile anesthetics on neuromuscular transmission is: desflurane > sevoflurane > isoflurane, depending on their blood-gas and tissue-gas solubility index.

Magnesium given intravenously during volatile anesthesia induces effects on neuromuscular transmission similar to that of neuromuscular blocking agents. This effect has never been investigated and quantified systematically and prospectively.

Propofol, an intravenous anesthetic, has very little effects on neuromuscular transmission. Therefore magnesium given intravenously during total intravenous anesthesia with propofol has no or only very little effect on neuromuscular transmission.

The primary objective of the study is to quantify the effect of a perfusion of intravenous magnesium on neuromuscular transmission measured by accelerometry with theTetraGraph device in patients undergoing general anesthesia with volatile anesthetics (desflurane, sevoflurane and isoflurane) as compared to intravenous anesthesia with propofol. The investigators expect a following rank order of the effect: desflurane > sevoflurane > isoflurane > propofol.

ELIGIBILITY:
Inclusion Criteria:

* Patients, age 18 to 65 years inclusive
* American Society of Anesthesiology [ASA] status I or II
* Body mass index 19 - 30 kg/m2
* Patient scheduled for elective surgery lasting ≥ 60 minutes
* Patient is able to read and understand the information sheet and to sign and date the consent form.
* Negative urinary or serum pregnancy test (not applicable if status post hysterectomy or tubal ligation or menopausal woman)

Exclusion Criteria:

* Surgery with need for neuromuscular block
* Contraindication for general anesthesia with laryngeal mask airway, such as gastro-oesophageal reflux.
* Hypersensitivity or allergy to magnesium sulfate or propofol
* Contraindication to volatile anesthetics such as malignant hyperthermia
* Patients with neuromuscular disease
* Patients receiving medications known to influence neuromuscular function (for instance, aminoglycosides or phenytoine)
* Known electrolyte abnormalities (for instance, hypermagnesemia)
* Atrioventricular heart block
* Patients with magnesium treatment within 48 hours before start of study
* Liver insufficiency (bilirubine <1.5x, ALAT/ASAT<2.5x the upper limit of normal value)
* Renal insuffisancy (créatinine <1.5x upper limit of normal value, clearance<30ml/minute)
* Patient having participated in any clinical trial within 30 days, inclusive, of signing the informed consent form of the current trial.
* Pregnant or breast-feeding women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 96 (Estimated)
Dates: Start 2022-11-18 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in TOF ratio after perfusion of magnesium | After starting TOF AUTO mode. patients will receive an intravenous perfusion of magnesium 60mg/kg mg kg-1 over 5 minutes. Neuromuscular monitoring will be continued until the end of surgery, but at least until a TOF ratio of 0.9 is reached.
  This primary outcome will be assessed with neuromuscular monitoring, carried out according to international guidelines. The ulnar nerve will be stimulated by train-of-four (TOF) using a TofScan monitor.

SECONDARY OUTCOMES:
Lowest T1 twitch height and TOF ratio | After the perfusion of magnesium and until the T1 twitch height and the TOF ratio reach the initial values again.
  The secondary outcomes are the lowest T1 twitch height and TOF ratio measured after starting the magnesium perfusion and the time required for the return of single twitch height (T1) and TOF ratio to its control value according to the TofScan measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Intensive Care, Valais Hospital, Sion, Switzerland

IPD SHARING:
Plan to Share IPD: No